CLINICAL TRIAL: NCT06600425
Title: A Phase 1b, Single-Center, Open-Label Study to Assess the Safety, Tolerability, Ciliary Rescue, and Pharmacodynamics of RCT1100 in Adults With Primary Ciliary Dyskinesia Caused by Pathogenic Mutations in the DNAI1 Gene
Brief Title: A Study to Assess the Safety, Tolerability, Ciliary Rescue, and Pharmacodynamics of RCT1100 in Adults With PCD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ReCode Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCT1100-102
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: Primary Ciliary Dyskinesia; PCD; Kartagener Syndrome
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PCD Participants (Experimental): RCT1100 mRNA therapy supplied to eligible participants with with Primary Ciliary Dyskinesia caused by disease-causing mutations in the DNAI1 gene
  Interventions: Drug: RCT1100

INTERVENTIONS:
Drug: RCT1100 — RCT1100 mRNA therapy supplied as varying dose strengths administered via oral inhalation using nebulizer

SUMMARY:
This is the second in-human study with RCT1100 and is designed to provide safety, tolerability and preliminary efficacy data for future clinical studies.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety, tolerability, ciliary rescue, pharmacodynamic biomarkers, and preliminary efficacy of RCT1100 following multiple doses of inhaled RCT1100 administered via nebulizer to participants with Primary Ciliary Dyskinesia caused by disease-causing mutations in the DNAI1 gene.

ELIGIBILITY:
Major Inclusion Criteria:

* Healthy, adult, male or female of, 18-70 years of age, inclusive, at screening.
* Participant has clinical diagnosis of PCD and disease-causing mutations in the DNAI1 gene
* Participant has a forced expiratory volume in one second (FEV1) of at least 50% predicted.

Major Exclusion Criteria:

* History or presence of clinically significant medical, surgical, clinical laboratory, or psychiatric condition or disease.
* History of cancer, with exception of adequately treated basal cell or squamous cell carcinoma of the skin.
* Predisposition to bleeding or clinically meaningful hemorrhagic event in the 12 months prior
* Medically significant hemoptysis.
* Anticoagulation therapy for the treatment of a pulmonary embolus or has had a pulmonary embolus in the last 6 months of screening.
* Active tuberculosis infection.
* 12-lead ECG with QT interval >450 msec (or >480 msec for BBB)
* Laboratory abnormalities in clinical laboratory tests at screening:

  1. Serum creatinine level
  2. Total bilirubin, aspartate aminotransferase or alanine aminotransferase values
  3. Hematological or coagulation values outside the normal reference range
* Any medical history of disease that has the potential to cause a rise in total bilirubin over the ULN.
* COVID-19 infection within 4 weeks of Screening or receipt of COVID-19 vaccine within 2 weeks prior to first dose of RCT1100.
* Receipt of vaccine with live virus, attenuated live virus, or live viral components within 2 weeks prior to first dose of RCT1100 or to receive these vaccines during treatment or within 8 weeks of completion of study treatment.

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
The number of participants with Adverse Events (AEs), including treatment-emergent adverse events (TEAEs) and Serious Adverse Events (SAEs). | From Baseline Through Week 24
  Safety and tolerability as assessed by number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs), as well as an adverse event of special interest (AESI): "Fever", which will include body temperature and any associated symptoms (chills, myalgia).

CONTACTS AND LOCATIONS:
Overall Officials: John Matthews, MBBS, MCRP, PhD, Study Chair — ReCode Therapeutics, Inc.; Michael Loebinger, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal Brompton Hospital, London
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No